CLINICAL TRIAL: NCT02576158
Title: HPV（Human Papillomavirus） Integration Testing for Cervical Cancer Screening
Brief Title: HPV Integration Testing for Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ding Ma, Chief Physician, Huazhong University of Science and Technology
Other Study IDs: CCS-01
Record Dates: First submitted 2015-09-22; First posted 2015-10-15 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Subjects will be women, 30-65 years of age: Patients who are at average risk of developing cervical intraepithelial neoplasia or cervical cancer who are eligible for cervical cancer screening will be asked to collect Cervical Exfoliated Cells sample for the HPV integration screening test and for the HPV testing and TCT. Subjects with HPV positive will undergo colposcopy within 90 days of enrollment.
  Interventions: Procedure: TCT，HPV，colposcopic inspection

INTERVENTIONS:
Procedure: TCT，HPV，colposcopic inspection

SUMMARY:
The primary objective is to determine the sensitivity and specificity of the HPV Integration-based cervical screening for detection of high-grade cervical intraepithelial neoplasia (CIN), using colposcopic inspection as the reference method. Lesions will be confirmed as malignant or CIN by colposcopic inspection and histopathologic examination.

ELIGIBILITY:
Inclusion Criteria:

Women aged 30-65 years old Attending the China population-based organised cervical screening program

Exclusion Criteria:

1. Not providing informed consent
2. previously confirmed CIN, cervical cancer, or other malignancies
3. previous therapeutic procedure to cervix
4. pregnancy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy women between the ages of 30 and 65 years
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-09 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
the sensitivity and specificity of the HPV Integration-based cervical screening for detection of high-grade cervical intraepithelial neoplasia (CIN)with comparison to HPV testing or TCT | 14 Months

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China